CLINICAL TRIAL: NCT03372980
Title: A Registry Study on Biomarkers of Takayasu's Arteritis
Brief Title: A Registry Study on Biomarkers of Takayasu's Arteritis (ARSBTA)
Status: Recruiting | Type: Observational
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ARSBTA
Record Dates: First submitted 2017-12-04; First posted 2017-12-14 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Takayasu's Arteritis
Keywords: Biomarkers
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood samples，Cells，Tissues
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case
- Control

SUMMARY:
Takayasu arteritis is a chronic vasculitis mainly involving the aorta and its main branches such as the brachiocephalic, carotid, subclavian, vertebral, and renal arteries, as well as the coronary and pulmonary arteries. Inflammation causes segments of the vessels to become narrowed, blocked, or even stretched, possibly resulting in aneurysms. The disease is very rare but most commonly occurs in young Asian women. However, there is a considerable lack of understanding of the disease mechanism of Takayasu arteritis. Initially, the disease remains clinically silent (or remains undetected) until the patients present with vascular occlusion. Additionally, many individuals with Takayasu arteritis, however, have no apparent symptoms despite disease activity. Therefore, biomarkers for diagnosis and monitor disease activity in individuals with Takayasu arteritis are needed. In this study, the investigators therefore to use different methods to identify new biomarkers for diagnosing or monitoring the disease activity in individuals with Takayasu arteritis. These biomarkers may provide valuable insights into the underlying biochemical processes and aid the understanding of the pathophysiology of this disease.

ELIGIBILITY:
Retrospective

Inclusion Criteria:

Subjects who met the American College of Rheumatology 1990 classification criteria for Takayasu arteritis:

1. Age of onset ≤40 years,
2. Claudication of upper or lower extremities,
3. Decreased pulsation of 1 or both brachial arteries,
4. Difference of ≥ 10 mmHg in systolic blood pressure between arms,
5. Bruit over subclavian arteries or aorta,
6. *Arteriographic evidence showing a branch of the aorta stenosis or occlusion.

Meeting more than 3 of 6 criteria suggests the diagnosis of Takayasu arteritis.

*Angiography in this study was replaced by vascular magnetic resonance angiography(MRA)or computed tomography angiography(CTA).

Exclusion Criteria:

1. Arteriographic lesions that could be entirely due to atherosclerosis,
2. Suffer from other autoimmune diseases (eg, ANCA-associated vasculitis, systemic lupus erythematosus, etc.) besides Takayasu arteritis,
3. Cogan's syndrome,
4. Behcet's disease,
5. Subjects with any serious acute or chronic infection,
6. Giant cell arteritis (large vessel vasculitis and at least 50 years old) or other infectious forms of large vessel vasculitis.

Prospective

Inclusion Criteria:

Subjects with initial suspicion of having Takayasu arteritis or patients with Takayasu arteritis need assessment of disease activity were prospectively enrolled.

Exclusion Criteria:

1. Patients without image studies.
2. Patients with confirmed other autoimmune diseases (eg, ANCA-associated vasculitis, systemic lupus erythematosus, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Case group consists of patients who was diagnosed as Takayasu's Arteritis; control group is general population without Takayasu's Arteritis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of each participant | These data is collected from the cases' medical record in an average of 3 month after the sample recruiting.
  Participant with Takayasu arteritis had image information from vascular magnetic resonance angiography (MRA) or computed tomography angiography (CTA) to confirm the final diagnosis.
Disease activity of each participant | These data is collected from the cases' medical record or during follow-up visit in an average of 6 month after the sample recruiting.
  Criteria for Disease Activity：Criteria for active disease are detection of new vascular lesion or lesions in arteries on vascular Imaging in participants who had undergone magnetic resonance angiography (MRA) or computed tomography angiography (CTA) examination in the month before evaluation, or at least 2 of the following: 1) new onset of carotodynia or pain over large vessels, 2) transient ischemic episodes not attributable to other factors, 3) new bruit or new asymmetry in pulses or blood pressure determination, 4) ischemic symptoms (including new-onset claudication), and 5) fever in absence of infection.
  Criteria defined inactive disease: 1) absence of the features of active disease for at least the previous 3 months; 2) absence of new vascular lesions and stability or improvement of previous vascular lesion or lesions on an imaging study performed up to 1 month before evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China